CLINICAL TRIAL: NCT06714838
Title: Rituximab Induced Remission in Patients With Chronic Inflammatory Demyelinating Polyneuropathy
Acronym: ReCIX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amsterdam University Medical Center (UMC), Location Academic Medical Center (AMC) (Other)
Collaborators: Stichting Treatmeds (Unknown); UMC Utrecht (Other); Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Filip Eftimov, Principal Investigator, MD PHD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024.0794; 2024-512506-25-00 (EU CTIS Number)
Record Dates: First submitted 2024-11-04; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: CIDP
Keywords: rituximab; remission; IVIg
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Rituximab

STUDY DESIGN:
Intervention Model Description: All patients will receive the same therapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm: all patients receive rituximab (Experimental): All patients will receive rituximab at baseline (1000 mg) and after two weeks (1000 mg). Then, depending of whether the patient shows improvement in the following three to six months, the patient will receive another dose of rituximab (500 mg) at six months.
  Interventions: Drug: Rituximab (Mabthera)

INTERVENTIONS:
Drug: Rituximab (Mabthera) — Rituximab will be administered in a hospital setting in the course of one day. It will be given intravenously, at time points baseline, week 2 and week 26.

SUMMARY:
The goal of this clinical trial is to learn if the drug called rituximab causes remission in patients with chronic inflammatory demyelinating polyneuropathy (CIDP). The aim is to investigate this in two types of patients, those who are newly diagnosed, and those who are already being treated and are dependent on the current standard therapy: immunoglobulins administered through infusion (IVIg) or through injection (SCIg). The main questions this trial aims to answer are:

* To assess the effectiveness of rituximab
* Whether it is possible and useful to prescribe patients rituximab who experience a relapse after at least six months after their last rituximab treatment.

Participants will:

* Receive the drug rituximab twice at the beginning of the trial and one additional time at six months.
* The newly diagnosed patients will also start another treatment called IVIg, which a nurse will administer every three weeks during the first three to six months.
* The patients who already being treated, will continue their regular treatment, until this is slowly reduced and stopped, during months three to six.
* Visit the clinic over the course of two years, during which they will have approximately 10 visits, for checkups and tests.
* Be asked to fill in questionnaires at each visit, and be asked to have their blood drawn four times.

DETAILED DESCRIPTION:
Rationale For almost 30 years, CIDP treatment consists of intravenous immunoglobulins (IVIg), corticosteroids or plasma exchange. Unfortunately, both IVIg and corticosteroids are considered treatments that suppress the disease rather than cure the disease, meaning that most patients starting on IVIg will require long-term maintenance treatment to avoid a relapse. Discovery of pathogenic antibodies in some patients with CIDP and the undisputed efficacy of anti- CD20 therapy in other demyelinating diseases such as multiple sclerosis has provided new arguments to introduce anti-CD20 therapy (such as rituximab) as a treatment modality in CIDP. In addition, rituximab (RTX) if now often used for/in treatment refractory CIDP cases and a recent review of retrospective studies has suggested efficacy in this group of patients. However, RTX efficacy data on new patients starting IVIg or patients who are on maintenance IVIg treatment is largely lacking. As RTX treatment has shown to lead to long-term remission in various auto-immune diseases, the hypothesis is that RTX can prevent ongoing need of IVIg treatment in CIDP.

Objective The primary objective of this study is to assess whether adding RTX to a limited period of IVIg induction treatment leads to long-term remission and discontinuation of IVIg, reducing the inconvenience of regular Ig infusions and related health care costs. Other objectives are to explore the feasibility of introducing rituximab as alternative maintenance treatment in patients with CIDP in patients who experience a relapse after at least 6 months after last RTX treatment (long term follow-up).

Main trial endpoints The investigators will include two groups of patients, namely untreated patients (Group 1) and immunoglobulin (Ig)-dependent patients (Group 2, see below, trial population). Primary outcome for both Group 1 and 2 is remission at 52 weeks after start of RTX. For Group 1, remission is defined as sustained improvement, without the need for further treatment. Improvement will be defined as decrease in disability by at least the minimal clinical important difference (MCID) on the adjusted INCAT (aINCAT) disability scale and/or the Inflammatory-Rasch Overall Disability Scale (IRODS).

Sustained is defined as no deterioration after maximal improvement achieved in week 13 to 26. For Group 2, remission is defined as no change in disability (MCID) between start of Ig withdrawal and week 52. Patients will be considered as a treatment failure if they do not meet the criteria for remission, or if they receive any immunomodulatory treatment for CIDP except RTX after discontinuation of induction treatment (Group 1), or withdrawal of maintenance Ig treatment (Group 2).

Other trial endpoints These will include various impairment measures, pain, fatigue, quality of life and adverse events. Endpoints will be assessed at 52 and 104 weeks, or earlier if a preliminary endpoint (relapse) is reached within the first year.

Trial design Multicentre, observational single arm study where patients will be participating for two years, including a 52 week intervention period and another 52 weeks for follow-up.

Trial population The study population will consist of two patient groups. In the first group (Group 1) new patients will be included, who are starting IVIg induction treatment. In the second group (Group 2) patients will be included who are already on maintenance IVIg or subcutaneous Ig (SCIg) treatment, and who are likely to be Ig dependent. Ig dependency will be defined as having wear-off symptoms before next IVIg infusion or SCIg administration suggesting active disease, patients with a documented failed IVIg/SCIg withdrawal attempt in the last year, or who required recent increase of IVIg/SCIg Protocol synopsis version 1.2, d.d. 15-07-2024 dosage with objective improvement.

Interventions Both groups will receive RTX, consisting of two infusion of 1000 mg per day two weeks apart (baseline) and a single infusion of 500 mg at 6 months. Because treatment effect of RTX can only be expected after 2-3 months, patients from Group 1 will initially receive concomitant IVIg induction treatment which will be stopped after 3-4 months. In Group 2, Ig will be tapered after 12 weeks by 25% during 3 infusions (IVIg) or in 2 months (SCIg). RTX will be administered at the hospital, as well as the first dose of IVIg of Group 1 (standard treatment), after which the IVIg can be administered at home.

Ethical considerations This study is considered of moderate risk. Side effects associated with RTX are well documented, and most often include infusion related reactions such as fever, hypertension, rash, tachycardia and fatigue and a moderately increased chance of infections The side effects associated with the combination of RTX and IVIg have not been previously studied in CIDP, however, these individual drugs have been studied extensively, and there is plenty of experience of combining these drugs in clinical practices in conditions such as myasthenia gravis, myositis and encephalitis. Therefore, the investigators do not expect unforeseen adverse events. For Group 2, there is a risk of a relapse if RTX does not lead to remission, in which case IVIg/SCIg will need to be restarted. Regular IVIg/SCIg withdrawals to assess Ig dependency are however part of standard care. Total follow-up of the study is 104 weeks. Follow-up hospital visits will be scheduled at 2, 8, 13, 26, 39, 52, 78 and 104 weeks. Unscheduled visits (including visits during relapses) can be scheduled at any time. For Group 1, potential benefits are related to the initial combination of IVIg and RTX: fast improvement and long-term remission, and possibly a higher proportion of patients improving as not all patients respond to IVIg. For Group 2, potential benefit is a long-term remission, thereby avoiding regular IVIg/SCIg infusions, associated side effects and high health care costs.

ELIGIBILITY:
Inclusion Criteria Group 1 (new/untreated patients):

* CIDP according to the EAN/PNS criteria (1)
* Untreated
* Men and women aged between 18 and 80 years
* Sufficient CIDP-related disability, as judged by treating physician to warrant IVIg and RTX treatment
* Capable of giving signed informed consent

Inclusion Criteria Group 2 (patients on maintenance treatment):

* CIDP according to the European association of neurology/Peripheral nerve society (EAN/PNS) criteria (1) on maintenance treatment (stable dose/interval of at least 4 infusions or 3 months), including one of the following categories:

  1. patients with wear-off symptoms before next IVIg infusion captured by at least the minimal clinical important difference (MCID) on at least one outcome measure (see below)
  2. patients with a failed withdrawal attempt in the last 12 months captured by at least an MCID on at least one outcome measure (see below)
  3. patients with an increase of IVIg/SCIg dose/interval in the last 12 months leading to improvement by at least the MCID on at least one outcome measure, see below.

     The most commonly used MCID criteria, namely: 1) one point on the aINCAT disability score (1-10); 2) 4 points on a centile score on I-RODS (disability, 1-100); 3) 2 points on the MRC sum score (muscle strength, 0-60) and 4) 8 kPa on Vigorimeter (grip strength, single or both arms, variable range).
* Men and women aged between 18 and 80 years
* Capable of giving signed informed consent

Exclusion Criteria:

* Paranodopathy with demonstrated (paranodal) antibodies, previously considered part of CIDP spectrum (in these cases rituximab is preferred treatment)
* Use of drugs associated with a demyelinating neuropathy in the last six months.
* Known serious adverse events with previous IVIg or RTX treatment. Hypersensitivity to RTX or any component of the formulation. Hypersensitivity to the human immunoglobulins or to any of the excipients. Known selective IgA deficiency patients who developed antibodies to IgA.
* Positive hepatitis B and C serology suggesting active/untreated infection (HBsAg, anti-HB core en anti-HBs and HCV antibody (IgG))
* Ongoing immunosuppressive treatment for other indications.
* Immunosuppressive treatment other than (already discontinued) corticosteroids in last 6 months.
* IVIg interval of once every 6 weeks or more than 6 weeks (applies to Group 2 only)
* Obesity (BMI > 35)
* Known active malignancy (not in remission), currently treated with chemotherapy or immunomodulatory drugs, or with a life expectancy of less than 1 year.
* History of recurrent/chronic infections
* Active, severe infections (such as tuberculosis, sepsis and opportunistic infections)
* Patients in a severely immunocompromised state Severe heart failure (New York Heart Association Class IV) or severe, uncontrolled cardiac disease
* Serious co-morbidity as judged by treating physician.
* Pregnancy or nursing mother; intention to become pregnant during the course of the study; female patients of childbearing potential either not using or not willing to use a medically reliable method of contraception for the entire duration of the study.
* No written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Remission at 52 weeks | Baseline to 52 weeks
  In order to assess efficacy of RTX:
  Remission at 52 weeks after start of RTX, i.e., no need of additional treatment after RTX treatment. For Group 1, remission is defined as sustained improvement, without the need for further treatment. Improvement will be defined as decrease in disability by at least the minimal clinical important difference (MCID) on the adjusted INCAT (aINCAT) disability scale and/or the Inflammatory-Rasch Overall Disability Scale (I-RODS). Sustained is defined as no deterioration after maximal improvement achieved in week 13 to 26. For Group 2, remission is defined as no change in disability (MCID) between start of Ig withdrawal and week 52.

OTHER OUTCOMES:
Stability on treatment at 104 weeks of follow-up. | Baseline to 104 weeks
  Explore the feasibility of introducing rituximab as alternative maintenance treatment in patients with CIDP in patients who experience a relapse after at least 6 months after last RTX treatment (long term follow-up):
  Definition for stability is similar to the primary outcome for Group 2, which is remission, defined as no change in disability (MCID) between weeks 52 and 104.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
As cidp is a rare disease, sharing of deidentified data will be considered in case of reasonable requests after publication of results.